CLINICAL TRIAL: NCT01284504
Title: The Effect Of Celecoxib On The Perioperative Inflammatory Response In Colon Cancer Patients - A Double-Blind Placebo-Controlled Trial
Brief Title: Effect of Celecoxib on Perioperative Inflammatory Response in Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual rate; the only participant withdrew after signing consent
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-19588; SU-10182010-7110 (Other: SU directory); COL0001 (Other: OnCore)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer; Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Experimental): Celecoxib, 200 mg tab
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): placebo, tab
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Celecoxib — 200 mg tablet oral
  Other Names: Celebrex; Celebra; Onsenal
  Arms: Celecoxib
Other: placebo — Placebo, tab
  Arms: Placebo

SUMMARY:
The proposed study aims to investigate how the administration of a drug known to reduce inflammation in humans, Celecoxib, will effect the peri-operative inflammatory response of a patient undergoing primary tumor resection surgery for colon cancer. The proposed project is an exploratory study, and will use data from blood samples and tumor samples to attempt to elucidate the immune and inflammatory response in colon cancer patients undergoing primary resection of their tumors.

DETAILED DESCRIPTION:
This study is the first to assess the perioperative time course of systemic inflammation and immunity in colon cancer patients and evaluate the effect of anti-inflammatory treatment with celecoxib on this response. In addition, evaluation of the effect of short-term preoperative administration of celecoxib on tumor immunogenicity will help us to understand how tumor-enhancing inflammation and anti-tumor immunity can be differentially affected by COX-2 inhibitors. The knowledge gained as a result of this research will help us to set up the infrastructure for a method to monitor the immunoinflammatory status of colon cancer patients with a longer term goal of designing interventions to suppress tumor-enhancing inflammation and vitalize anti-tumor immunity in the perioperative period. The long-term objective is to use these novel tools in order to improve cancer-specific survival in patients with colon cancer after primary tumor resection.

ELIGIBILITY:
Inclusion Criteria:

- Colon cancer patients with no evidence of metastasis in distant organs (i.e., TNM stage I-III), who are

* between 18 and 75 years old,
* have a body mass index (BMI) between 18 and 35 kg/m^2,
* and are eligible for laparoscopically-assisted colectomy for primary tumor resection.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

- A history of allergic-type reactions to celecoxib or sulphonamides,

* a history of asthma, skin reactions or other allergic reactions to aspirin or other NSAIDs,
* a history of thromboembolic event (cerebrovascular accident, transient ischemic attack,
* unstable angina, myocardial infarction, deep vein thrombosis, or pulmonary embolism),
* renal insufficiency (defined by a serum creatinine level > 1.5 mg/dL or blood urea nitrogen level > 22 mg/dL),
* active gastrointestinal bleeding in the 60 days before surgery,
* alcohol or drug abuse, and
* previous chemotherapy or abdominal/pelvic radiation therapy.
* After randomization, other exclusion criteria will include a surgical procedure longer than 6 h, inability to extubate the trachea within 4 h after operation, evidence of a new postoperative myocardial infarction, abnormal postoperative mental status or any new neurologic deficit, significant postoperative bleeding (with a hemoglobin level < 7.5 g/dL), requiring blood transfusion, or a urine output of less than 30 mL/h.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 patient was consented but withdrew before treatment assignment (randomization), none were treated.
Groups:
- Celocoxib: Celecoxib: 200 mg tablet oral
- Placebo: placebo
  placebo
Period: Overall Study
Arm/Group | Celocoxib | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Sample - Analyzed for TCR Repertoire and Global Transcription Profiling
Time Frame: 2 years
Population: One patient was accrued and withdrawn after signing consent; none were treated.
Arm/Group | Celocoxib | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Blood Samples Taken Before Initiation of Study, Day of Surgery, Days 1 and 3 Post-op, and 30 Days Post-op. Analyzed for 50 Serum Cytokines, Cell-specific Gene Expression, and TCR Repertoire.
Time Frame: 30 days
Population: One patient was accrued and withdrawn after signing consent; none were treated.
Arm/Group | Celocoxib | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Surveys to Evaluate Patient Pain, Fatigue, and Quality of Recovery, Recorded From Day of Surgery to 30 Days Post-op.
Time Frame: 30 days
Population: One patient was accrued and withdrawn after signing consent; none were treated.
Arm/Group | Celocoxib | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Celecoxib | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No